CLINICAL TRIAL: NCT04973137
Title: A Phase 3, Randomized, Multicenter, Double-Blind, Placebo-Controlled, Efficacy and Safety Study of Birtamimab Plus Standard of Care vs. Placebo Plus Standard of Care in Mayo Stage IV Subjects With Light Chain (AL) Amyloidosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Birtamimab in Mayo Stage IV Patients With AL Amyloidosis
Acronym: AFFIRM-AL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The AFFIRM-AL clinical trial did not meet its primary endpoint.
Sponsor: Prothena Biosciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEOD001-301
Record Dates: First submitted 2021-07-01; First posted 2021-07-22 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-07

CONDITIONS: Light Chain (AL) Amyloidosis
Keywords: Light Chain (AL) Amyloidosis; Mayo Stage IV; birtamimab
MeSH Terms: conditions — Amyloidosis | interventions — birtamimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Birtamimab plus Standard of Care Chemotherapy- For Double-blind Phase and OLE Phase of study (Experimental): Intravenous administration of 24 mg/kg birtamimab every 28 days.
  Drug: Standard of Care Chemotherapy. Bortezomib-containing chemotherapy regimen (e.g. cyclophosphamide, bortezomib, and dexamethasone (CyBorD)) according to the institutional standard of care.
  The initiation of daratumumab treatment at randomization is allowed at the discretion of the Investigator; initiation at any other time during the Double-blind Phase is prohibited. For subjects who did not initiate daratumumab at randomization during the Double-blind Phase, daratumumab may be initiated at any time during the OLE Phase at the Investigator's discretion.
  Interventions: Drug: Birtamimab; Drug: Standard of Care Chemotherapy
- Placebo plus Standard of Care Chemotherapy- For Double-blind Phase of study (Placebo Comparator): Intravenous 0.9% Saline administration as a placebo every 28 days.
  Drug: Standard of Care Chemotherapy. Bortezomib-containing chemotherapy regimen (e.g. cyclophosphamide, bortezomib, and dexamethasone (CyBorD)) according to the institutional standard of care. Initiation of daratumumab at randomization allowed at the discretion of the investigator.
  Interventions: Other: Placebo; Drug: Standard of Care Chemotherapy

INTERVENTIONS:
Drug: Birtamimab — Intravenous administration of 24 mg/kg birtamimab every 28 days
  Arms: Birtamimab plus Standard of Care Chemotherapy- For Double-blind Phase and OLE Phase of study
Other: Placebo — Intravenous 0.9% Saline administration as a placebo every 28 days
  Arms: Placebo plus Standard of Care Chemotherapy- For Double-blind Phase of study
Drug: Standard of Care Chemotherapy — Bortezomib-containing chemotherapy regimen (e.g. cyclophosphamide, bortezomib, and dexamethasone (CyBorD)) according to the institutional standard of care

SUMMARY:
A Phase 3 study to evaluate the efficacy and safety of birtamimab plus standard of care compared to placebo plus standard of care in Mayo Stage IV patients with AL amyloidosis.

DETAILED DESCRIPTION:
This is a Phase 3 multicenter, global, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of birtamimab in Mayo Stage IV patients with AL amyloidosis (i.e., Double-blind Phase), followed by a long-term, open-label extension (i.e., Open-label Extension [OLE] Phase). The primary objective of the Double-blind Phase is to evaluate the efficacy of birtamimab by assessing time to all-cause mortality. All patients will receive bortezomib-containing chemotherapy regimen as standard of care.

For the Double-blind Phase of the study, approximately 220 newly diagnosed Mayo Stage IV patients with AL amyloidosis will be enrolled and randomized in a 2:1 ratio to birtamimab or placebo. Subjects will remain on study until study completion, when the pre-defined number of events (all-cause mortality) have been reached.

After completion of the Double-blind Phase, eligible subjects may enter the optional OLE Phase, in which all subjects will receive open-label birtamimab treatment, regardless of Double-blind Phase randomized treatment assignment. Treatment in the OLE Phase will continue for an additional 24 months or until birtamimab is commercially available in a subject's country of residence, whichever occurs first (in accordance with country-specific regulations). The primary objective of the OLE Phase is to evaluate the long-term safety of birtamimab plus standard of care in Mayo Stage IV subjects with AL amyloidosis.

ELIGIBILITY:
Key Inclusion Criteria for Double-blind Phase:

* Aged ≥18 years and legal age of consent according to local regulations
* Newly diagnosed and AL amyloidosis treatment-naïve with cardiac involvement
* Confirmed diagnosis of AL amyloidosis
* Confirmed Mayo Stage IV AL Amyloidosis as defined by NT-proBNP ≥1800 pg/mL and Troponin-T ≥0.025 ng/mL or high sensitivity cardiac troponin T≥40ng/L and dFLC ≥18 mg/dL
* Planned first-line chemotherapy contains bortezomib administered subcutaneously weekly

Inclusion Criteria for Open-label (OLE) Phase:

* Must not have discontinued treatment in Double-blind Phase
* WOCBP must have a negative pregnancy test and must agree to use highly effective contraception through 90 days following last study drug administration
* Male subjects must be surgically sterile or agree to use highly effective contraception through 90 days following last study drug administration
* Ability to understand and willingness to sign an ICF prior to initiating the OLE Phase

Key Exclusion Criteria for Double-blind Phase:

* Non-AL amyloidosis
* NT-proBNP >8500 pg/mL
* Meets the International Myeloma Working Group (IMWG) definition of multiple myeloma except for malignancy biomarker of involved/uninvolved serum free light chain ratio ≥100
* Subject is eligible for and plans to undergo ASCT or organ transplant during the study
* Myocardial infarction, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or ECG evidence of acute ischemia, within 6 months prior to the Month 1-Day 1 Visit
* Severe valvular stenosis (e.g., aortic or mitral stenosis with a valve area <1.0 cm2) or severe congenital heart disease
* ECG evidence of acute ischemia or active conduction system abnormalities
* Prior treatment with hematopoietic growth factors, transfusions of blood or blood products within 1 week of Month 1-Day 1
* Prior radiotherapy within 4 weeks of Month 1-Day 1
* Prior treatment with plasma cell-directed chemotherapy, birtamimab, daratumumab, 11- 1F4, anti-serum amyloid P antibody, doxycycline for amyloid, or other investigational treatment directed at amyloid
* Waldenström's macroglobulinemia and/or immunoglobulin M monoclonal gammopathy

Exclusion Criteria for OLE Phase:

* Any medical condition or clinically significant abnormality on physical, neurological, laboratory, vital signs, or ECG examination that precludes treatment with birtamimab or participation in the study, in the medical judgment of the Investigator
* Symptomatic orthostatic hypotension that in the medical judgment of the Investigator would interfere with subject's ability to safely receive treatment or complete study assessments
* History of Grade ≥3 infusion-related AEs during the Double-blind Phase or hypersensitivity to birtamimab
* Unable or unwilling to adhere to the study-specified procedures and restrictions
* Planning to use any other investigational treatment during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (110):
- United States (22):
  - Yale Cancer Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Trumbull, Trumbull, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - Johns Hopkins University, Bethesda, Maryland
  - Boston University School of Med., Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Perlmutter Cancer Center - 38th Street, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - New York University Langone Hospital - Long Island, New York, New York
  - Duke Clinical Research Institute, Durham, North Carolina
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - The Ohio State University College of Medicine, Columbus, Ohio
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt - Ingram Cancer Center - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - University of Washington, Seattle, Washington
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - SESLHD: St George Hospital, Kogarah, New South Wales
  - Royal Perth Hospital, Perth, Western Australia
- Austria (4):
  - Paracelsus Medical University, Salzburg, Salzburg
  - Paracelsus Medical University, Salzburg
  - Medizinische Universität Wien, Vienna
  - Medizinische Universität, Vienna
- Belgium (4):
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Ostend, Oostende
  - Centre Hospitalier Universitaire Universite Catholique de Louvain - Site Godinne, Yvoir, Yvoir
  - AZ Sint-Jan Brugge-Oostende AV, Ostend
  - CHU UCL Namur (Site Godinne), Yvoir
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Royal Victoria Hospital, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice ostrava, Ostrava-Poruba, Moravian-Silesian
  - Všeobecná fakultní nemocnice v Praze, Prague, Prague
- Odense Universitetshospital, Odense, Region Syddanmark, Denmark
- France (13):
  - Hôpital Bretonneau, Tours, Centre-Val de Loire
  - Hôpitaux Universitaires Henri Mondor, Créteil, Créteil
  - Hôpital Haut-Lévêque, Pessac, Gironde
  - Pitie-Salpêtrière Hospital, Paris, Ill-de-France
  - Hopital Necker, Paris, Ill-de-France
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Lorraine
  - Hopital Rangueil, Toulouse, Midi-Pyrenees
  - Hôpital Claude Huriez, Lille, Nord
  - CHU Nantes, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire Poitiers, Poitiers, Vienne
  - CHU de Bordeaux, Bordeaux
  - Hopital Henri Mondor, Creteil, Créteil
  - Hôpital Necker-Enfants Malades, Paris
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Uniklinik Köln, Köln, Baden-Wurttemberg
  - University Medicine Mainz, Mainz, Rhineland-Palatinate
- Greece (3):
  - Alexandra General Hospital, Athens, Attica
  - Theagenio Anti-Cancer Hospital of Thessaloniki, Thessaloniki, Central Macedonia
  - University Hospital of Patras, Patra, Peloponnese
- Semmelweis Egyetem - I. sz. Belgyógyászati Klinika, Budapest, Budapest, Hungary
- Ireland (2):
  - Cork University Hospital, Cork, Munster
  - Cancer Clinical Trials and Research Unit, Beaumont Hospital, Dublin
- Israel (6):
  - Bnai Zion Medical Center, Haifa, Haifa District
  - Rambam Medical Center, Haifa, Haifa District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Ashkelon, Southern District
  - Barzilai Medical Center, Ashkelon
  - Carmel Medical Center, Haifa
- Italy (2):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
- Japan (6):
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Kyoto Kuramaguchi Medical Center, Kita, Kyoto
  - Shinshu University Hospital, Matsumoto, Nagano
  - Jichi medical university hospital, Shimotsuke, Tochigi
  - Red Cross Medical Center, Shibuya-ku, Tokyo
  - Nagoya City University Hospital, Aichi
- Netherlands (2):
  - Maastricht Universitair Medisch Centrum, Maastricht, Limburg
  - Universitair Medisch Centrum Groningen, Groningen, Provincie Groningen
- Klinika Hematologii i Transplantologii, Gdansk, Pomeranian Voivodeship, Poland
- Portugal (2):
  - Hospital de Braga, Braga, Braga District
  - Centro Hospitalar Universitário Lisboa Norte - Hospital De Santa Maria, Lisbon, Lisbon District
- South Korea (9):
  - Keimyung University Dongsan Hospital, Daegu, Gyeongsangbuk-do
  - Chonnam National University Hwasun Hospital, Gwangju, Jeollanam-do
  - Samsung Medical Center, Seoul, Seoul
  - Severance Hospital, Seoul, Seoul Teugbyeols
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea - Seoul St. Mary's Hospital, Seoul
- Spain (12):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Català d'Oncologia - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clinic of Barcelona, Barcelona, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals, Barcelona, Barcelona
  - University Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Josep Trueta ICO Girona, Girona, Girona
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Clinica Universidad de Navarra -Madrid, Pamplona, Navarre
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital Universitario 12 de Octubre, Vila-real
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital, Taipei City, Taipei
  - Taipei Veterans General Hospital, Taipei, Taipei
- Turkey (Türkiye) (4):
  - Ankara UMF, Ankara, Ankara
  - Gazi University, Ankara, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir, İzmir
- United Kingdom (4):
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, High Heaton, England
  - Barts Health NHS Trust, London, England
  - University College London Hospitals, London, England
  - Manchester University NHS Foundation Trust, Manchester, England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gertz MA, Cohen AD, Comenzo RL, Kastritis E, Landau HJ, Libby EN, Liedtke M, Sanchorawala V, Schonland S, Wechalekar A, Zonder JA, Palladini G, Walling J, Guthrie S, Nie C, Karp C, Jin Y, Kinney GG, Merlini G. Birtamimab plus standard of care in light-chain amyloidosis: the phase 3 randomized placebo-controlled VITAL trial. Blood. 2023 Oct 5;142(14):1208-1218. doi: 10.1182/blood.2022019406. PMID 37366170

RESULTS

PARTICIPANT FLOW:
Groups:
- Birtamimab (24 mg/kg) + Standard of Care: Double Blind Phase: Birtamimab, 24 mg/kg IV every 4 weeks with Standard of Care
  Open Label Extension Phase: Birtamimab, 24 mg/kg IV every 4 weeks with Standard of Care
- Placebo + Standard of Care: Double Blind Phase: Placebo 0.9% Saline IV every 4 weeks with Standard of Care
  Open Label Extension Phase: Birtamimab, 24 mg/kg IV every 4 weeks with Standard of Care
Period: Double Blind Phase
Arm/Group | Birtamimab (24 mg/kg) + Standard of Care | Placebo + Standard of Care
Started (Participants randomized and dosed) | 139 | 68
Completed | 97 | 49
Not Completed | 42 | 19
Not completed — Adverse Event | 4 | 0
Not completed — Death | 25 | 15
Not completed — Physician Decision | 5 | 1
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Other | 2 | 2
Period: Open Label Extension Phase
Arm/Group | Birtamimab (24 mg/kg) + Standard of Care | Placebo + Standard of Care
Started (Not all double-blind participants enrolled in Open-Label Extension) | 92 | 44
Completed | 0 | 0
Not Completed | 92 | 44
Not completed — Death | 3 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study Terminated by Sponsor | 83 | 43
Not completed — Site Terminated by Sponsor | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Birtamimab (24 mg/kg) + Standard of Care: Birtamimab, 24 mg/kg IV every 4 weeks with Standard of Care
- Placebo + Standard of Care: Placebo 0.9% Saline IV every 4 weeks with Standard of Care
- Total: Total of all reporting groups
Arm/Group | Birtamimab (24 mg/kg) + Standard of Care | Placebo + Standard of Care | Total
Number analyzed (Participants) | 139 | 68 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 31 | 84
  >=65 years | 86 | 37 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (10.38) | 64.1 (8.88) | 65.2 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 24 | 77
  Male | 86 | 44 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 27 | 13 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 99 | 44 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  Hungary | 0 | 1 | 1
  United States | 31 | 14 | 45
  Czechia | 0 | 2 | 2
  Japan | 7 | 2 | 9
  United Kingdom | 3 | 3 | 6
  Portugal | 1 | 0 | 1
  Spain | 13 | 6 | 19
  Greece | 10 | 4 | 14
  Canada | 7 | 1 | 8
  Austria | 3 | 3 | 6
  Netherlands | 7 | 4 | 11
  South Korea | 12 | 7 | 19
  Turkey | 1 | 3 | 4
  Belgium | 1 | 0 | 1
  Taiwan | 4 | 2 | 6
  Italy | 3 | 1 | 4
  Israel | 5 | 1 | 6
  Australia | 3 | 3 | 6
  France | 21 | 8 | 29
  Germany | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 121 | 62 | 183
  Unknown or Not Reported | 15 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Time to All-cause Mortality for the Double Blind Phase
Description: Comparison of time to all-cause mortality for birtamimab and placebo control.
Time Frame: Time from the first dose of study drug until the pre-defined number of events (all-cause mortality) have been reached, assessed up to 39 months.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Birtamimab (24 mg/kg) + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 139 | 68
Participants
  Event (Death) Occurred | 32 | 17
  Number of Subjects Censored | 107 | 51
Statistical Analysis 1: Comparison: Birtamimab (24 mg/kg) + Standard of Care; Test type: Superiority; p = 0.7680, Log Rank; Hazard Ratio (HR) = .915, 95% CI 2-sided [.508 to 1.649]

2. Secondary Outcome: 6MWT Distance at Month 9
Description: Change from baseline to Month 9 in the 6-Minute Walk Test (6MWT) distance calculated as the value at 9 months minus the value at baseline.
Time Frame: Month 9
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: Meters
Arm/Group | Birtamimab (24 mg/kg) + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 139 | 68
Meters | 4.5 [-52.00 to 50.50] | 7.75 [-33.00 to 36.00]
Statistical Analysis 1: Comparison: Birtamimab (24 mg/kg) + Standard of Care; Test type: Superiority; p = 0.5288, Rank ANCOVA; Hodge-Lehmann Median Difference (Net) = -8.50, 95% CI 2-sided [-35.47 to 18.46]

3. Secondary Outcome: Physical Component Summary Score of the Short Form-36, Version 2 at Month 9
Description: Change from baseline to Month 9 in the Short Form-36, version 2 (SF-36) calculated as the value at 9 months minus the value at baseline.
  SF-36 v2 is a 36-item self-administered quality-of-life questionnaire that measures health on functional status, well-being, and overall evaluation of health. The Physical Component Summary score ranges from 0 to 100 with higher scores indicating higher health-related quality of life. The Physical Component Summary is derived primarily from questions regarding physical functioning, physical problems, bodily pain, and general health questions.
Time Frame: Month 9
Population: ITT Population
Measure: Median (Inter-Quartile Range); unit: Score
Arm/Group | Birtamimab (24 mg/kg) + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 139 | 68
Score | 1.710 [-2.695 to 6.920] | 4.205 [-0.430 to 10.320]
Statistical Analysis 1: Comparison: Birtamimab (24 mg/kg) + Standard of Care; Test type: Superiority; p = 0.9597, Rank ANCOVA; Hodge-Lehmann Median Difference (Net) = 0.34, 95% CI 2-sided [-2.68 to 3.37]

ADVERSE EVENTS:
Time Frame: Initiation of study drug through the last study visit or up to 28 days after last dose, whichever is later, assessed up to 39 months.
Description: Safety Analysis Set included all participants who received at least one dose of study drug.
Groups:
- Birtamimab (24 mg/kg) + Standard of Care (Double-Blind Phase): Birtamimab, 24 mg/kg IV every 4 weeks with Standard of Care in Double-Blind Phase
- Placebo + Standard of Care (Double-Blind Phase): Placebo 0.9% Saline IV every 4 weeks with Standard of Care in Double-Blind Phase
- Birtamimab (24 mg/kg) + Standard of Care (Open Label Extension Phase): Birtamimab, 24 mg/kg IV every 4 weeks with Standard of Care in Open Label Extension Phase
Arm/Group | Birtamimab (24 mg/kg) + Standard of Care (Double-Blind Phase) | Placebo + Standard of Care (Double-Blind Phase) | Birtamimab (24 mg/kg) + Standard of Care (Open Label Extension Phase)
All-Cause Mortality (participants affected / at risk) | 32/139 | 17/68 | 3/136
Serious Adverse Events (participants affected / at risk) | 83/139 | 39/68 | 17/136
Other Adverse Events (participants affected / at risk) | 136/139 | 66/68 | 53/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Birtamimab (24 mg/kg) + Standard of Care (Double-Blind Phase) (N=139) | Placebo + Standard of Care (Double-Blind Phase) (N=68) | Birtamimab (24 mg/kg) + Standard of Care (Open Label Extension Phase) (N=136)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 27 | 14 | 3
Cardiac arrest (Cardiac disorders) | 5 | 5 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 6 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Ulcerative gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Sudden death (General disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 2 | 1 | 0
Cardiac death (General disorders) | 2 | 0 | 0
Chills (General disorders) | 2 | 0 | 0
Generalised oedema (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0
ABO incompatibility (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 3 | 2
COVID-19 (Infections and infestations) | 2 | 4 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Septic shock (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 1 | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Disseminated varicella zoster virus infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumococcal infection (Infections and infestations) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0
Scrotal infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 2
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Troponin T increased (Investigations) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 4 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 8 | 4 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Birtamimab (24 mg/kg) + Standard of Care (Double-Blind Phase) (N=139) | Placebo + Standard of Care (Double-Blind Phase) (N=68) | Birtamimab (24 mg/kg) + Standard of Care (Open Label Extension Phase) (N=136)
Anaemia (Blood and lymphatic system disorders) | 34 | 16 | 3
Neutropenia (Blood and lymphatic system disorders) | 11 | 6 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 5 | 0
Cardiac failure (Cardiac disorders) | 19 | 7 | 1
Atrial fibrillation (Cardiac disorders) | 14 | 5 | 0
Angina pectoris (Cardiac disorders) | 0 | 5 | 0
Dry eye (Eye disorders) | 7 | 4 | 0
Constipation (Gastrointestinal disorders) | 49 | 24 | 0
Diarrhoea (Gastrointestinal disorders) | 40 | 20 | 4
Nausea (Gastrointestinal disorders) | 38 | 25 | 0
Vomiting (Gastrointestinal disorders) | 20 | 6 | 1
Abdominal distension (Gastrointestinal disorders) | 20 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 9 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 7 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 7 | 3 | 0
Acquired macroglossia (Gastrointestinal disorders) | 7 | 2 | 1
Ascites (Gastrointestinal disorders) | 7 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4 | 0
Oedema peripheral (General disorders) | 41 | 24 | 4
Fatigue (General disorders) | 24 | 13 | 1
Pyrexia (General disorders) | 19 | 7 | 1
Asthenia (General disorders) | 17 | 4 | 1
Chills (General disorders) | 11 | 3 | 1
Influenza like illness (General disorders) | 7 | 4 | 1
Oedema (General disorders) | 7 | 4 | 1
Localised oedema (General disorders) | 7 | 1 | 0
Non-cardiac chest pain (General disorders) | 6 | 4 | 1
Hypogammaglobulinaemia (Immune system disorders) | 9 | 3 | 0
COVID-19 (Infections and infestations) | 19 | 7 | 0
Urinary tract infection (Infections and infestations) | 15 | 8 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 9 | 2
Nasopharyngitis (Infections and infestations) | 11 | 6 | 2
Respiratory tract infection (Infections and infestations) | 8 | 4 | 1
Pneumonia (Infections and infestations) | 7 | 5 | 0
Bronchitis (Infections and infestations) | 7 | 3 | 1
Hordeolum (Infections and infestations) | 7 | 3 | 1
Herpes zoster (Infections and infestations) | 0 | 4 | 0
Fall (Injury, poisoning and procedural complications) | 8 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 7 | 3 | 2
Lymphocyte count decreased (Investigations) | 18 | 12 | 3
Weight decreased (Investigations) | 15 | 8 | 1
Aspartate aminotransferase increased (Investigations) | 14 | 2 | 0
Blood creatinine increased (Investigations) | 13 | 8 | 0
Alanine aminotransferase increased (Investigations) | 13 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 11 | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 9 | 4 | 1
Platelet count decreased (Investigations) | 7 | 4 | 1
White blood cell count decreased (Investigations) | 7 | 3 | 1
Neutrophil count decreased (Investigations) | 7 | 2 | 1
Weight increased (Investigations) | 5 | 5 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 26 | 12 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 21 | 6 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 12 | 4 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 14 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 4 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 24 | 8 | 0
Dizziness (Nervous system disorders) | 22 | 10 | 3
Dysgeusia (Nervous system disorders) | 18 | 3 | 0
Headache (Nervous system disorders) | 16 | 5 | 2
Neuropathy peripheral (Nervous system disorders) | 9 | 5 | 0
Syncope (Nervous system disorders) | 8 | 6 | 0
Tremor (Nervous system disorders) | 3 | 4 | 0
Insomnia (Psychiatric disorders) | 22 | 13 | 2
Anxiety (Psychiatric disorders) | 8 | 5 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 4 | 0
Chronic kidney disease (Renal and urinary disorders) | 6 | 4 | 1
Haematuria (Renal and urinary disorders) | 6 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 12 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 14 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 7 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 4 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 11 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 7 | 0
Hypotension (Vascular disorders) | 22 | 14 | 2
Orthostatic hypotension (Vascular disorders) | 11 | 5 | 0
Hypertension (Vascular disorders) | 7 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT04973137/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT04973137/SAP_001.pdf